CLINICAL TRIAL: NCT05267860
Title: The Efficacy and Safety of Using Prophylactic Abdominal Drainage After Cholecystectomy: A Randomized Control Trial.
Brief Title: The Efficacy and Safety of Using Prophylactic Abdominal Drainage After Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aleppo (Other)
Responsible Party: Principal Investigator, Ahmad Yamen Arnaout, Principal Investigator, University of Aleppo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Drainage After Cholecystectomy
Record Dates: First submitted 2022-02-21; First posted 2022-03-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Drainage; Laparoscopic Cholecystectomy; Acute Cholecystitis
Keywords: Prophylactic Drainage; Laparoscopic cholecystectomy; Acute cholecystitis.; Upper GI Surgery; Cholecystitis; Choledocholithiasis; Gallbladder Diseases
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis; Choledocholithiasis; Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with a prophylactic drain after cholecystectomy (Experimental)
  Interventions: Device: Prophylactic Drain
- Patients without using any prophylactic Drainage after cholecystectomy (No Intervention)

INTERVENTIONS:
Device: Prophylactic Drain — We want to put a prophylactic drain after cholecystectomy.
  Arms: Patients with a prophylactic drain after cholecystectomy

SUMMARY:
Investigators want to assess the safety and efficacy of using abdominal drainage with not using any drainage, by estimating different outcomes after laparoscopic cholecystectomy for different reasons. Patients are seen at the Accident and Emergency Department or in the surgical wards at Aleppo University Hospital (AUH) over 12 months period.

DETAILED DESCRIPTION:
The routine use of prophylactic drainage has become common in many hospitals around the world after cholecystectomy for different reasons. In elective surgeries, the evidence does not support the use of drainage. But in emergency laparoscopic cholecystectomy surgeries, using drainage remains controversial. Surgeons who support the use of drainage find it useful to identify the early complications of surgery and removing intra-abdominal collections, while opponents of drainage use believe that it increases the risk of wound infection. But, a systematic review and meta-analysis discussed the ineffectiveness of the routine use of the prophylactic drainage after laparoscopic cholecystectomy for acute cholecystitis and requested more randomized clinical trial studies on the subject. However, this study and others in the medical literature contain very few high-quality randomized controlled trials, hence our randomized controlled trial compares the use and non-use of drainage in patients undergoing laparoscopic cholecystectomy for different reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients are seen at the Accident and Emergency Department or in the surgical wards at Aleppo University Hospital (AUH) over 12 months period.
* Patients who undergo cholecystectomy for any reason.

Exclusion Criteria:

* Non-cooperative patients for regular follow up.
* Draining for therapeutic indications.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Morbidity /Complications | 30 days after the operation
  overall complication rate; graded by the Clavien- Dindo complications classification system.

SECONDARY OUTCOMES:
Intraperitoneal abscess | up to 30 days
  The patient will be monitored and followed up for 30 days after the surgery, and the necessary investigations will be requested to diagnose if the patient has an Intraperitoneal abscess
Wound infection/ Surgical site infection | up to 30 days
  Surgical site infection has been defined and classified as superficial incisional, deep incisional, and organ/ space_ surgical site infection by the Centers for Disease Control and Prevention (CDC) (Anderson 2014; Ban 2017; Berríos-Torres 2017).

OTHER OUTCOMES:
Adverse events from the operation | up to 24 hours
Mortality | up to 30 days
Hospital stay | up to 30 days
  Number of days, patient in hospital since admission

CONTACTS AND LOCATIONS:
Locations (1):
- Aleppo University Hospital, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: Yes
We will publish the data after publishing the research.

REFERENCES:
- [Background] Antoniou S, Koch O, Antoniou G, Kohler G, Chalkiadakis G, Pointner R, Granderath F. Routine versus no drain placement after elective laparoscopic cholecystectomy: meta-analysis of randomized controlled trials. Minerva Chir. 2014 Jun;69(3):185-94. PMID 24970306
- [Background] Gurusamy KS, Koti R, Davidson BR. Routine abdominal drainage versus no abdominal drainage for uncomplicated laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2013 Sep 3;(9):CD006004. doi: 10.1002/14651858.CD006004.pub4. PMID 24000011
- [Background] Monson JR, Guillou PJ, Keane FB, Tanner WA, Brennan TG. Cholecystectomy is safer without drainage: the results of a prospective, randomized clinical trial. Surgery. 1991 Jun;109(6):740-6. PMID 2042093
- [Background] Wong CS, Cousins G, Duddy JC, Walsh SR. Intra-abdominal drainage for laparoscopic cholecystectomy: A systematic review and meta-analysis. Int J Surg. 2015 Nov;23(Pt A):87-96. doi: 10.1016/j.ijsu.2015.09.033. Epub 2015 Sep 18. PMID 26386402
- [Derived] Arnaout AY, Kadoura L, Masri R, Nerabani Y, Atli AA, Arnaout K, Arnaout I, Bsata A, Kayali H, Mahli N, Al-Haj A, Ayoub K, Niazi A, Ghazal A; Aleppo University Hospital Team. The efficacy and safety of using prophylactic abdominal drainage after laparoscopic cholecystectomy: A randomized control trial. Health Sci Rep. 2024 Aug 8;7(8):e2284. doi: 10.1002/hsr2.2284. eCollection 2024 Aug. PMID 39131596